CLINICAL TRIAL: NCT06915272
Title: Effects of Head and Neck Cooling on Environmental Symptom Management and Mood in People With Multiple Sclerosis During Sailing
Brief Title: Effects of Sailing and Cooing in the Quality of Life of Multiple Sclerosis Individuals
Acronym: MS Sailing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Antonia Kaltsatou, PhD, Adjunct Assistant Professor in Clinical Exercise Physiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1300
Record Dates: First submitted 2025-03-17; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cooling Intervention (Experimental): Head and Neck Cooling Intervention
  Interventions: Other: Head and Neck Cooling Intervention
- Control (No Intervention)

INTERVENTIONS:
Other: Head and Neck Cooling Intervention — Participants received a head and neck cooling intervention involving the daily use (≥2 hours/day) of cooling devices consisting of a cooling cap and cooling towel specifically designed for localized head and neck cooling. Devices were activated by immersing them in cold water maintained at approximately 10°C.
  Arms: Cooling Intervention

SUMMARY:
In this study, we aim to evaluate the impact of head and neck cooling on symptoms and psychological states in individuals with Multiple Sclerosis (MS) during a 7-day Oceans of Hope Challenge sailing trip around the Greek islands of the Argosaronic Gulf in May 2023. Forty-five individuals with relapsing-remitting MS will participate in the sailing trip. Participants will be allocated to either a Cooling group (n=25), using a cooling cap and neck towel for at least two hours per day, or a Control group (n=20) without cooling interventions.

Before and after the trip, participants will complete the Functional Assessment of Multiple Sclerosis Scale (FAMS), the Environmental Symptoms Questionnaire (ESQ), and the abbreviated 40-item Profile of Mood States (POMS-40). These assessments will be used to evaluate quality of life, environmental symptoms, and mood states.

The study is designed to examine whether daily use of head and neck cooling during a prolonged outdoor activity influences MS-related symptoms, quality of life, and psychological well-being.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic neurodegenerative disease characterized by physical and cognitive impairments that significantly affect patients' quality of life. Common symptoms include fatigue, mobility limitations, cognitive difficulties, anxiety, depression, and social isolation. Exercise is widely recognized as beneficial for managing MS symptoms; however, participation in structured exercise programs remains low due to barriers such as fear, negative past experiences, or lack of interest.

This study aims to explore whether unstructured outdoor leisure activities, specifically sailing combined with head and neck cooling, can help reduce symptom severity and improve psychological states in individuals with MS. Outdoor leisure activities have demonstrated positive effects on psychological and emotional health by reducing depression, improving mood, and promoting social engagement. Sailing, which combines physical activity and social interaction, may enhance quality of life in people with MS. However, sensitivity to increases in body temperature is a known challenge for individuals with MS, as it can exacerbate symptoms and deter physical activity participation. Cooling strategies, such as head and neck cooling, have been used to help maintain thermal comfort and support symptom management.

The objective of this study is to assess the impact of daily head and neck cooling on MS symptoms and psychological well-being during a 7-day sailing trip (Oceans of Hope Challenge) in the Argosaronic Islands, Greece. Ethical approval was obtained from the Greek Multiple Sclerosis Society.

A total of 45 participants with relapsing-remitting MS will be randomly assigned to either a Cooling group or a Control group. The Cooling group will use head and neck cooling devices daily for a minimum of two hours during the sailing trip, while the Control group will participate without cooling interventions. Both groups will engage in daily sailing activities, navigation tasks, and island exploration.

Participants will complete three questionnaires before and after the trip: the Functional Assessment of MS Scale (FAMS) to assess quality of life, the Environmental Symptoms Questionnaire (ESQ-IV) to evaluate general well-being and symptom severity, and the Profile of Mood States (POMS-40) to assess mood states.

Statistical analyses will include two-way repeated measures ANOVA and independent t-tests to evaluate within- and between-group differences over time. The study is designed to determine whether integrating cooling strategies into outdoor leisure activities can reduce MS symptom severity, improve psychological well-being, and potentially encourage greater participation in therapeutic recreational activities.

ELIGIBILITY:
Inclusion Criteria: Were adults aged 18 years or older. Had a confirmed diagnosis of relapsing-remitting multiple sclerosis (RRMS) based on the 2017 McDonald criteria.

Had experienced no relapse within the past six months. Had an Expanded Disability Status Scale (EDSS) score between 0 and 5.5, indicating the ability to walk at least 100 meters independently without assistance.

Had a documented history of heat sensitivity confirmed by their physician. Had not used any cooling therapy within at least four months prior to study participation.

Were fluent in English (for accurate completion of questionnaires and instructions).

Exclusion Criteria: Used medications specifically prescribed to manage psychological MS-related symptoms (e.g., antidepressants, psychostimulants).

Had experienced an MS relapse within the past six months. Had an Expanded Disability Status Scale (EDSS) score greater than 5.5 (unable to walk at least 100 meters independently).

Had no documented history of heat sensitivity related to MS. Had used any cooling therapies within four months prior to the study participation.

Were unable to understand or communicate fluently in English.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-06 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Change in MS-related symptoms and heat sensitivity (as measured by Environmental Symptoms Questionnaire - ESQ-IV) | Change from baseline to immediately after the 7-day intervention period.
  Evaluated by comparing total symptom scores before and after the 7-day sailing intervention between the cooling group and the control group.
  This outcome directly assesses the effectiveness of the head and neck cooling intervention in managing MS symptoms exacerbated by heat stress.

SECONDARY OUTCOMES:
Change in Mood Disturbances | Change from baseline to immediately after the 7-day intervention period.
  The Profile of Mood States (POMS-40) will be used to assess mood disturbances across several dimensions, including tension, depression, confusion, anger, vigor, and fatigue.

OTHER OUTCOMES:
Change in Quality of Life Assessed by the Functional Assessment of Multiple Sclerosis (FAMS) Total Score | Change from baseline to immediately after the 7-day intervention period.
  The Functional Assessment of MS Scale (FAMS) will be used to assess quality of life across the following domains: mobility, MS-related symptoms, emotional well-being, general contentment, thinking/fatigue, and family/social well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Kaltsatou, PhD, Principal Investigator — Department of Physical Education and Sport Science, University of Thessaly
Locations (1):
- Greek Multiple Sclerosis Society, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to protect participant confidentiality and privacy, as the informed consent obtained did not include provisions for data sharing with third-party researchers.